CLINICAL TRIAL: NCT03508258
Title: Investigating the Association of Type of Anticoagulation Treatment for Non-valvular Atrial Fibrillation and Risk of Bleeding in England
Brief Title: Study to Describe Risk of Bleeding in Patients Depending on the Different Anticoagulant Therapy They Are on for Atrial Fibrillation (AF)
Status: Withdrawn | Type: Observational
Why Stopped: Study was discontinued in 2018 as sufficient sample size was not met.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-664
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with NVAF starting Apixaban
  Interventions: Other: Non-interventional
- Participants with NVAF starting Warfarin
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional
  Groups: Participants with NVAF starting Apixaban
Other: Non-Interventional — Non-Interventional
  Groups: Participants with NVAF starting Warfarin

SUMMARY:
Study of patients with nonvalvular atrial fibrillation (NVAF) who are newly prescribed NOACs (Novel Oral Anticoagulants) in routine clinical practice in England

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atrial fibrillation at or prior to index (the initiation of treatment)
* Incident prescription of an oral anticoagulant (index date)
* Patients with at least one year of computerized data prior to index date

Exclusion Criteria:

* Patients identified with a diagnosis of mechanical heart valve replacement or mitral stenosis identified at any point in the pre-index period in either CPRD by Read codes or in HES as ICD-10/OPCS codes
* Patients with indication of venous thromboembolism (pulmonary embolism or deep vein thrombosis) identified in in either CPRD by Read codes or HES by ICD-10/OPCS codes within 3 months prior to index

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF patients newly prescribed NOACs in England
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding | At the end of 1 year
Incidence of intracranial bleeding | At the end of 1 year
Incidence of gastrointestinal bleeding | At the end of 1 year
Incidence of clinically relevant non-major bleeding | At the end of 1 year
Incidence of ischemic stroke | At the end of 1 year
Incidence of unspecified stroke | At the end of 1 year
Incidence of systemic embolic events | At the end of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Bethesda, Maryland, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm